CLINICAL TRIAL: NCT00966394
Title: Changes in Salivary Bacteria and Oral Health Status in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Salivary Bacteria and Oral Health Status in Children With ADHD
Acronym: ADHD
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Moti Moskovitz, Department of Pediatric Dentistry, Hadassah School of Dental Medicine
Other Study IDs: adhd-hmo-ctil
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2009-08

CONDITIONS: Attention Deficit Hyperactivity Disorders; Caries, Dental; Xerostomia
Keywords: ADHD, saliva, caries
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dental Caries; Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ADHD medication: Children with ADHD and pharmacologic treatment
- ADHD without medication: Children with ADHD without pharmacologic treatment
- healthy: Healthy children ASA1

SUMMARY:
Attention deficit and hyperactivity (ADHD) affect 6% of school-aged children. Few studies reported higher prevalence of caries and restorations among children with ADHD. Methylphenidate is the drug of choice to treat ADHD. according to the medical literature methylphenidate can cause xerostomia.

Our study will investigate saliva parameters (such as quantity, bacteria in saliva, buffer capacity), oral hygiene and diet habits and their influence on caries among children with ADHD and among healthy children.

Our hypothesis is:

* Children with ADHD will have more caries.
* Children with ADHD will have more detrimental oral hygiene and diet habits.
* There will be a difference in the saliva parameters between children with ADHD and healthy children.

ELIGIBILITY:
Inclusion Criteria:

* test group- diagnosis of ADHD.
* control group- ASA1

Exclusion Criteria:

* control group
* administration of medicine at the time of the check-up.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with ADHD, treated by medications or not, treated in the neurologic clinic at Hadassah.
  The control are healthy children visiting the pediatric dental clinic at Hadassah.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah school of dental medicine, Jerusalem, Israel